CLINICAL TRIAL: NCT04085653
Title: Managed Access Program (MAP) Cohort Treatment Plan CBYL719F12001M to Provide Access to Alpelisib (BYL719) for Patients With PIK3CA-Related Overgrowth Spectrum (PROS)
Brief Title: Managed Access Program (MAP) to Provide Access to Alpelisib (BYL719) for Patients With PIK3CA-Related Overgrowth Spectrum (PROS)
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719F12001M; NCT04473040 (obsolete NCT alias)
Record Dates: First submitted 2019-09-05; First posted 2019-09-11 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: PIK3CA-Related Overgrowth Spectrum (PROS)
Keywords: adult; pediatric; BYL719; PIK3CA; Overgrowth Spectrum; PROS; alpelisib
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — Alpelisib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: alpelisib — Alpelisib will be provided as 50 mg, 125mg and 200 mg film coated tablets as individual patient supply, and will be dosed on a flat scale of mg/day not to be adjusted to body weight or surface area.
  In Adult patients, alpelisib will be administered at a starting dose of 250 mg orally once daily on a continuous dosing schedule and can be adjusted for toxicity per the recommendations in this treatment plan.
  In Pediatric patients, alpelisib will be administered at a maximum starting dose of 50 mg orally once daily on a continuous dosing schedule and can be interrupted for toxicity per the recommendations in this treatment plan; no dose reductions are allowed.
  Other Names: BYL719

SUMMARY:
The purpose of this Cohort Treatment Plan is to allow access to alpelisib for patients diagnosed with PIK3CA-Related Overgrowth Spectrum (PROS) who fulfill certain eligibility criteria as specified in this document. The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations

The US Expanded Access Program is closed.

ELIGIBILITY:
Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

1. Adult or pediatric patients with a diagnosis of PROS preferably with evidence of a mutation in the PIK3CA gene
2. The treating physician has determined that the patient's condition is severe or life threatening, treatment is necessary and there are no other feasible alternatives for the patient.
3. Confirmed adequate bone marrow function Written patient informed consent must be obtained prior to start of treatment

Exclusion criteria

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. Patient has history of hypersensitivity to any drugs or metabolites of PI3K inhibitor or any of the excipients of alpelisib.
2. Patient with uncontrolled diabetes mellitus type I or not controlled type II (based on fasting plasma glucose (FPG) and HbA1c)
3. Patient who has other concurrent severe and/or uncontrolled medical conditions that would, in the Treating Physician's judgment, contraindicate administration of alpelisib (eg. active or uncontrolled severe infection, chronic active hepatitis, immuno-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.)
4. Patient has a known history of Severe Cutaneous Adverse Reactions (SCAR) like Steven Johnson's syndrome (SJS), Erythema Multiforme (EM), Toxic Epidermal Necrolysis (TEN), or Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS).
5. History of pancreatitis within 1 year of screening or past medical history of chronic pancreatitis
6. Chronic liver disease patients with Child Pugh score B or C
7. Subjects with unresolved osteonecrosis of the jaw
8. Subject is currently receiving any of the following medications and cannot be discontinued 7 days prior to the start of the treatment:

   * Strong inducers of CYP3A4
   * Inhibitors of BCRP
9. Patient has a known history of Human Immunodeficiency Virus (HIV) infection (testing not mandatory unless required by local regulations or requirements).
10. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to start of program treatment, or who have not fully recovered from side effects of such treatment.

    Note: The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
11. Male patient who does not use highly effective contraception during the treatment with alpelisib and through the duration as defined below after the final dose of alpelisib. Sexually active males should use a condom during intercourse while taking drug and for at least 1 week after stopping alpelisib and should not father a child in this period. In addition, male participants must not donate sperm during study and up to the time period specified above.
12. Subject or caregiver (in the case of a pediatric subject) is not able to understand and to comply with treatment instructions and requirements
13. Subject is a nursing (lactating) or pregnant woman as confirmed by a positive serum (hCG) test prior to initiating study treatment
14. Subject is a woman of child-bearing potential defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during study treatment and at least for 1 week after the last dose of any study treatment.

Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptom-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least 6 weeks before taking study treatment. In case of unilateral oophorectomy, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject
* Use of oral (estrogen and progesterone), injected or implanted combined hormonal method of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormonal vaginal ring or transdermal hormone contraception. In case of use or oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Note: Women are considered postmenopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea and/or confirmed by hormonal status (FSH and estradiol) or have undergone surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least 6 weeks before taking study treatment. In the case of unilateral oophorectomy, only when the reproductive status of the woman had been confirmed by hormonal levels (FSH and estradiol), she will be considered not of child bearing potential

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult